CLINICAL TRIAL: NCT03366818
Title: Efficacy and Safety of VERSI System for Acute Ischemic Stroke
Brief Title: New Stent Retriever, VERSI System for AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kobe City General Hospital (Other)
Responsible Party: Principal Investigator, Nobuyuki Sakai, Director, Neurosurgery, Kobe City General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NEURO0001
Record Dates: First submitted 2017-11-11; First posted 2017-12-08 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thrombectomy (Experimental): thrombectomy by Versi system
  Interventions: Device: thrombectomy

INTERVENTIONS:
Device: thrombectomy — mechanical thrombectomy

SUMMARY:
To confirm efficacy and safety of VERSI system for acute ischemic stroke

DETAILED DESCRIPTION:
Efficacy; TICI 2a or more recanalization upto 3 pass of study device Safety; symptomatic intracranial hemorrhage within 24 hours of procedure

ELIGIBILITY:
Inclusion Criteria:

* onset to treat within 8 hours
* NIHSS 8 or more
* ASPECTS 5 or more
* Target vessel is ICA, MCA, VA, BA, PCA
* non-eligible or failed IV rt-PA

Exclusion Criteria:

* known hemorrhagic tendency
* arterial dissection, vasculitis
* allergy for contrast media
* other inappropriate condition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
incidence of treatment-related severe adverse event | within 24 hours after procedure
  symptomatic intracranial hemorrhage

SECONDARY OUTCOMES:
recovery to independent life {modified Rankin score of 2 or less] | 90days after procedure
  Proportion of subjects who have modified Rankin Scale (mRS) score of 2 or less
all intracralnial hemorrhage | within 24 hours after procedure
  incidence of symptomatic and asymptomatic intracranial hemorrhage
acceptable clinical outcome | 90days after procedure
  Proportion of subjects who have modified Rankin Scale (mRS) score of 2 or less or back to baseline of mRS
Severe adverse event related to device | within 24 hours after procedure
  Any severe adverse event related to device
recanalization ability of device | immediatry after procedure
  rate of immediate reperfusion with the device upto 3 path measured using Thrombolysis in Cerebrovascular Infarction (TICI) score of 2b or greater

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sakai, MD DMSc, Principal Investigator — Kobe City Medical Center General Hospital, Kobe, Japan
Locations (1):
- Kobe City General Hospital, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakai N, Imamura H, Adachi H, Tani S, Tokunaga S, Funatsu T, Suzuki K, Adachi H, Sasaki N, Kawabata S, Akiyama R, Horiuchi K, Ohara N, Kono T, Fujiwara S, Kaneko N, Tateshima S. First-in-man experience of the Versi Retriever in acute ischemic stroke. J Neurointerv Surg. 2019 Mar;11(3):296-299. doi: 10.1136/neurintsurg-2018-014040. Epub 2018 Sep 27. PMID 30262657